CLINICAL TRIAL: NCT04389398
Title: A Randomized, Controlled Study of Preventing Effects of Pocket Hematoma After Implantation Cardiovascular Implanted Electronic Devices With Pocket Compression Fixation Belt
Brief Title: Prevention of Pocket Hematoma After Implantation Cardiovascular Implanted Electronic Devices
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: XJTU1AF2020LSK-040
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Hematoma Postoperative; Cardiac Resynchronization Therapy Devices; Compression Bandages

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pocket compression fixation belt (Experimental): Pocket compression belt is used to compress the bleeding vessels and reduce bleeding after implantation.
  Interventions: Device: pocket compression fixation belt
- Sand bag compression (Active Comparator): Sand bag compression is used to compress the bleeding vessels and reduce bleeding after implantation.
  Interventions: Device: pocket compression fixation belt

INTERVENTIONS:
Device: pocket compression fixation belt — Pocket compression fixation belt to is used to compress the postoperative wounds of CIEDS patients, and its effect of preventing hematoma is evaluated.

SUMMARY:
As the number of implanted cardiovascular implanted electronic devices (CIEDs) increases, the incidence of their complications also grows. Pocket hematoma is an important complication of CIED implantation, which has been reported in 2.9-9.5% of CIEDs patients. Pocket hematoma can cause significant pain and interfere with proper wound healing, and it also increased the risk of infection and may prolong length of stay.

Pocket compression is usually applied to compress bleeding vessels and reduce bleeding after implantation. A conventional compression method is to place a sandbag over the pocket, and then using adhesive tape to fix the sandbag. Due to adhesive tape is elastic and the tape may be pulled by patients' activity, sandbag easily migrated from the site. Therefore, nurse must readjust the position of sandbag, or even remove the adhesive tape and perform re-compress. Furthermore, adhesive tape can cause skin erosion. All of which not only result in patients' discomfort and dissatisfaction, but also increase the burden on nurses and wastes resources.

We designed a pocket compression fixation belt. We assumed that using this fixation belt can ensure the compression effect while avoiding sand bag displacement, reducing skin erosion and decrease the workload of care.

ELIGIBILITY:
Inclusion Criteria:

* Registry of patients undergoing PM, ICD, and CRT-P or CRT-D device implantation in The First Affiliated Hospital of Xi'an Jiaotong University.

Exclusion Criteria:

* (1) age<18 years or >80 years, (2) a history of any psychiatric illness, (3) a history of open wounds in the infraclavicular region, (4) coagulation disorder or bleeding diathesis, (5) anticoagulation or antithrombotic treatments could not be interrupted, (6) refusing to participate. This study was approved by the Ethics Committee of the First Affiliated Hospital of Xi'an Jiaotong University (approval number XJTU1AF2020LSK-040).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-05-25 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
The incidence and grade of pocket hematoma | 48 hours post implantation of ICEDs.
  The incidence and grade of pocket hematoma between the control and experimental group were compared

SECONDARY OUTCOMES:
Operation time and positional adjustment of the sandbag | Accumulate the time used to place and adjust the salt bag within 48 hours for each patient.
  Operation time refer to the consuming minutes that perform compression procedure for each patient, including the total time to fix the salt bag and remove the salt bag twice during intermittent compression.

CONTACTS AND LOCATIONS:
Overall Officials: Jingwen Hu, Master, Study Chair — First Affiliated Hospital Xi'an Jiaotong University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Epstein AE, DiMarco JP, Ellenbogen KA, Estes NA 3rd, Freedman RA, Gettes LS, Gillinov AM, Gregoratos G, Hammill SC, Hayes DL, Hlatky MA, Newby LK, Page RL, Schoenfeld MH, Silka MJ, Stevenson LW, Sweeney MO, Tracy CM, Epstein AE, Darbar D, DiMarco JP, Dunbar SB, Estes NA 3rd, Ferguson TB Jr, Hammill SC, Karasik PE, Link MS, Marine JE, Schoenfeld MH, Shanker AJ, Silka MJ, Stevenson LW, Stevenson WG, Varosy PD; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines; Heart Rhythm Society. 2012 ACCF/AHA/HRS focused update incorporated into the ACCF/AHA/HRS 2008 guidelines for device-based therapy of cardiac rhythm abnormalities: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2013 Jan 22;61(3):e6-75. doi: 10.1016/j.jacc.2012.11.007. Epub 2012 Dec 19. No abstract available. PMID 23265327
- [Background] European Society of Cardiology (ESC); European Heart Rhythm Association (EHRA); Brignole M, Auricchio A, Baron-Esquivias G, Bordachar P, Boriani G, Breithardt OA, Cleland J, Deharo JC, Delgado V, Elliott PM, Gorenek B, Israel CW, Leclercq C, Linde C, Mont L, Padeletti L, Sutton R, Vardas PE. 2013 ESC guidelines on cardiac pacing and cardiac resynchronization therapy: the task force on cardiac pacing and resynchronization therapy of the European Society of Cardiology (ESC). Developed in collaboration with the European Heart Rhythm Association (EHRA). Europace. 2013 Aug;15(8):1070-118. doi: 10.1093/europace/eut206. Epub 2013 Jun 24. No abstract available. PMID 23801827
- [Background] Kusumoto FM, Schoenfeld MH, Wilkoff BL, Berul CI, Birgersdotter-Green UM, Carrillo R, Cha YM, Clancy J, Deharo JC, Ellenbogen KA, Exner D, Hussein AA, Kennergren C, Krahn A, Lee R, Love CJ, Madden RA, Mazzetti HA, Moore JC, Parsonnet J, Patton KK, Rozner MA, Selzman KA, Shoda M, Srivathsan K, Strathmore NF, Swerdlow CD, Tompkins C, Wazni O. 2017 HRS expert consensus statement on cardiovascular implantable electronic device lead management and extraction. Heart Rhythm. 2017 Dec;14(12):e503-e551. doi: 10.1016/j.hrthm.2017.09.001. Epub 2017 Sep 15. No abstract available. PMID 28919379
- [Background] Raatikainen MJP, Arnar DO, Merkely B, Nielsen JC, Hindricks G, Heidbuchel H, Camm J. A Decade of Information on the Use of Cardiac Implantable Electronic Devices and Interventional Electrophysiological Procedures in the European Society of Cardiology Countries: 2017 Report from the European Heart Rhythm Association. Europace. 2017 Aug 1;19(suppl_2):ii1-ii90. doi: 10.1093/europace/eux258. PMID 28903470
- [Background] Sridhar AR, Yarlagadda V, Yeruva MR, Kanmanthareddy A, Vallakati A, Dawn B, Lakkireddy D. Impact of haematoma after pacemaker and CRT device implantation on hospitalization costs, length of stay, and mortality: a population-based study. Europace. 2015 Oct;17(10):1548-54. doi: 10.1093/europace/euv075. Epub 2015 Apr 7. PMID 25855676
- [Background] Palmisano P, Accogli M, Zaccaria M, Luzzi G, Nacci F, Anaclerio M, Favale S. Rate, causes, and impact on patient outcome of implantable device complications requiring surgical revision: large population survey from two centres in Italy. Europace. 2013 Apr;15(4):531-40. doi: 10.1093/europace/eus337. Epub 2013 Feb 13. PMID 23407627
- [Background] Sohail MR, Hussain S, Le KY, Dib C, Lohse CM, Friedman PA, Hayes DL, Uslan DZ, Wilson WR, Steckelberg JM, Baddour LM; Mayo Cardiovascular Infections Study Group. Risk factors associated with early- versus late-onset implantable cardioverter-defibrillator infections. J Interv Card Electrophysiol. 2011 Aug;31(2):171-83. doi: 10.1007/s10840-010-9537-x. Epub 2011 Mar 2. PMID 21365264
- [Background] Koh Y, Bingham NE, Law N, Le D, Mariani JA. Cardiac implantable electronic device hematomas: Risk factors and effect of prophylactic pressure bandaging. Pacing Clin Electrophysiol. 2017 Jul;40(7):857-867. doi: 10.1111/pace.13106. Epub 2017 Jun 14. PMID 28543543
- [Background] Baddour LM, Epstein AE, Erickson CC, Knight BP, Levison ME, Lockhart PB, Masoudi FA, Okum EJ, Wilson WR, Beerman LB, Bolger AF, Estes NA 3rd, Gewitz M, Newburger JW, Schron EB, Taubert KA; American Heart Association Rheumatic Fever, Endocarditis, and Kawasaki Disease Committee; Council on Cardiovascular Disease in Young; Council on Cardiovascular Surgery and Anesthesia; Council on Cardiovascular Nursing; Council on Clinical Cardiology; Interdisciplinary Council on Quality of Care; American Heart Association. Update on cardiovascular implantable electronic device infections and their management: a scientific statement from the American Heart Association. Circulation. 2010 Jan 26;121(3):458-77. doi: 10.1161/CIRCULATIONAHA.109.192665. Epub 2010 Jan 4. PMID 20048212
- [Derived] Hu J, Zheng J, Liu X, Li G, Xiao X. Effect of a pocket compression device on hematomas, skin reactions, and comfort in patients receiving a cardiovascular implantable electronic device: a randomized controlled trial. J Interv Card Electrophysiol. 2022 Mar;63(2):275-281. doi: 10.1007/s10840-021-00973-5. Epub 2021 Mar 6. PMID 33675448